CLINICAL TRIAL: NCT00838721
Title: Prospective Evaluation of the Efficacy of Pascal Trabeculoplasty: A Pilot Study
Brief Title: Evaluation of Pascal Laser Trabeculoplaty
Acronym: PLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Clara Valley Health & Hospital System (Other)
Collaborators: OptiMedica Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PASCAL-1
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2009-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Ocular Hypertension; Laser Trabeculoplasty
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laser trabeculoplasty — Deliver laser energy to the trabecular meshwork using the Pascal Laser System

SUMMARY:
Laser Trabeculoplasty has been shown to be effective in lowering intraocular pressure (IOP) in patients with primary open-angle glaucoma (POAG). Although initially demonstrated with the Argon laser (ALT), several other laser systems have also been employed with comparable efficacy. Recently, Selective Laser Trabeculoplasty (SLT) has been shown to lower intraocular pressure comparable to ALT. The advantage of SLT is that the target eye structure, the trabecular meshwork, remains intact with minimal damage at the cellular level. In contrast, ALT lowers IOP at the expense of scarring of the trabecular meshwork. The purpose of this study is to evaluate the efficacy of lowering IOP with Pascal Laser Trabeculoplasty (PLT) employing reduced energy levels compared to ALT and a computer guided pattern of laser treatment applications.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy males and females, older than 18 years of age with two (2) sighted eyes
2. Have OAG, PXG, or combined mechanism glaucoma - as long as their angles are open
3. Have uncontrolled IOP (>24mmHg); or controlled with Medicine(s)
4. If on medical treatment, have undergone a washout period of at least one month prior to Pascal treatment
5. Able and willing to comply with the treatment/follow-up schedule and requirements;
6. Able to provide written informed consent

Exclusion Criteria:

1. Pregnant, intending to become pregnant during course of study, less than 3 months postpartum or less than 6 weeks after completion of breastfeeding
2. Have an advanced visual field defect within 10° of fixation
3. Have had previous glaucoma surgery, except for peripheral iridotomy
4. Have corneal disease obviating the use of corneal applanation for a reliable IOP measurement, or would cause difficulty in viewing the TM by means of gonioscopic lens
5. Using systemic steroids
6. Participation in a study of another device or drug within 3 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria
7. Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study
8. No concomitant use of IOP lowering medicine (Group 1)
9. No co-existing ocular pathology with the exception of Cataract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | 1 week, 1 month, 3 months, 6 months, 9 months and 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Engelman, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, San Jose, California, United States